CLINICAL TRIAL: NCT01077544
Title: A Multi-center, Open-label, Pharmacokinetic Study of Oral Nilotinib in Pediatric Patients With Newly Diagnosed Chronic Phase (CP) Ph+ CML, With CP or Accelerated Phase (AP) Ph+ CML Resistant/Intolerant to Imatinib and/or Dasatinib, or With Refractory/Relapsed Ph+ ALL
Brief Title: A Pharmacokinetic (PK) Study of Nilotinib in Pediatric Patients With Philadelphia Chromosome-positive (Ph+) Chronic Myelogenous Leukemia (CML) or Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2120; 2010-018419-14 (EudraCT Number)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-10

CONDITIONS: Chronic Myeloid Leukemia; Acute Lymphoblastic Leukemia
Keywords: Chronic Myeloid Leukemia; Acute Lymphoblastic Leukemia; Ph+ CML; Ph+ ALL; pediatric; nilotinib; imatinib; chronic phase; accelerated phase; newly diagnosed Ph+ CML; dasatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): 1 year to < 10 years pediatric patients with newly diagnosed CP-Ph+ CML, or CP or AP-Ph+ CML resistant/intolerant to imatinib and/or dasatinib, or relapsed/refractory Ph+ ALL (acute lymphoblastic leukemia) treated at the proposed dose of 230 mg/m2 bid.
  Interventions: Drug: Nilotinib
- Group 2 (Experimental): >= 10 years to <18 years pediatric patients with newly diagnosed CP-Ph+ CML, or CP or AP-Ph+ CML resistant/intolerant to imatinib and/or dasatinib, or relapsed/refractory Ph+ ALL (acute lymphoblastic leukemia) treated at the proposed dose of 230 mg/m2 bid.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib capsules were delivered in bottles with dose strengths of 50mg, 150mg and 200mg.
  Patients were administered nilotinib 230 mg/m2 (per BSA) bid, orally, rounded to the nearest 50 mg (max single dose 400 mg) for 28 days (1 cycle) for up to 12 cycles prior to protocol amendment 3 and up to 24 cycles post amendment 3. Capsules were to be swallowed whole with water. Apple sauce (puréed apple) may have been used as a vehicle for dosing where capsules were not able to be swallowed whole with water.
  Other Names: AMN107

SUMMARY:
This study will assess the pharmacokinetics of nilotinib in Ph+ CML pediatric patients that are newly diagnosed or resistant or intolerant to imatinib or dasatinib or refractory or relapsed Ph+ ALL compared to the adult populations. It will also evaluate safety and activity of nilotinib as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Must have one of the following: newly diagnosed CP Ph+CML, CP or AP resistant/ intolerant to imatinib and/or dasatinib, or Ph+ ALL either relapsed after or refractory to standard therapy
* adequate renal, hepatic and pancreatic function

Exclusion Criteria:

* patients receiving therapy with strong CYP3A4 inhibitors and/or inducers and treatments cannot be stopped or changed to a different medication at least 14 days prior to starting study drug
* patients receiving therapy with any medications with a known risk or possible risk to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
* gastrointestinal impairment or disease that may interfere with drug absorption
* liver, pancreatic or severe renal disease unrelated to disease under study
* impaired cardiac function
* patients who received dasatinib within 3 days of starting study drug
* patients who received imatinib within 5 days of starting study drug
* patients receiving hydroxyurea or corticosteroids that has not been discontinued at least 1 week after initiation of nilotinib
* patients who received hematopoietic growth factors within 7 days of starting study drug or Pegfilgrastim (Neulasta®) within 14 days of starting study drug
* patients with Stem Cell Transplant (SCT) or Rescue without TBI: Evidence of active graft vs. host disease and < 3 months since SCT

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2011-04-14 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- France (4):
  - Novartis Investigative Site, Bordeaux, Aquitaine
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
- Italy (3):
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Roma, RM
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- United Kingdom (3):
  - Novartis Investigative Site, West Midlands, Birmingham
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Bristol

REFERENCES:
- See also: Results for CAMN107A2120 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14405

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 1 year to < 10 years pediatric patients
- Group 2: >= 10 years to <18 years pediatric patients
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 8 | 7
Completed | 5 | 2
Not Completed | 3 | 5
Not completed — New Cancer Therapy | 3 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): consists of all patients who passed the screening and are enrolled into the study. Patients may or may not have taken study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.8 (1.16) | 13.7 (2.81) | 10.0 (4.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 3 | 8
Weight [Mean (Standard Deviation); unit: kg] | 24.60 (4.739) | 48.89 (17.533) | 35.93 (17.328)
Height [Mean (Standard Deviation); unit: cm] | 119.9 (7.49) | 158.0 (16.32) | 137.7 (23.02)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 16.962 (1.7654) | 18.944 (3.4563) | 17.887 (2.7795)

OUTCOME MEASURES:

1. Primary Outcome: Summary of Nilotinib Non-compartmental PK Parameters: Cmax
Description: The full PK profiles of nilotinib in pediatric patients were assessed using serial sampling following a single 230 mg/m2 dose on Cycle 1 Day 1.
Time Frame: Cycle 1 Day 1
Population: Pharmacokinetic Analysis Set (PAS) consists of all patients who received the nilotinib dose on Day 1, had an evaluable Day 1 PK profile or provided at least one evaluable steady state trough concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 7
ng/mL | 405.111 (42.5) | 402.715 (35.2)

2. Secondary Outcome: Number of Ph+ CML Participants With Confirmed Complete Hematologic Response (CHR)
Description: A confirmed complete hematological response (CHR) is defined when all of the following criteria are achieved at two consecutive assessments, at least 4 weeks apart: white blood cell (WBC) count < 10 × 109/L; platelet < 450 × 109/L; basophils < 5%; no blasts and promyelocytes in peripheral blood (PB); myelocytes + metamyelocytes < 5% in PB; and no extramedullary involvement. The information used for hematological assessment was to be obtained from the laboratory and extramedullary data, all merged by patient and date.
Time Frame: minimum of 12 cycles (28 days per cycle)
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 6
Participants
  Yes | 5 | 5
  No | 0 | 1

3. Primary Outcome: Summary of Nilotinib Non-compartmental PK Parameters: Tmax
Description: as for outcome 1
Time Frame: Cycle 1 Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 7
h | 2.000 (163.1050) [1.02 to 7.08] | 3.000 (140.8314) [2.00 to 7.88]

4. Primary Outcome: Summary of Nilotinib Non-compartmental PK Parameters: AUClast (Last = 24h)
Description: as for outcome 1
Time Frame: Cycle 1 Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 7
ng*h/mL | 4160.969 (38.5) | 5707.368 (51.2)

5. Primary Outcome: Summary of Nilotinib Non-compartmental PK Parameters: AUC0-12h
Description: as for outcome 1
Time Frame: Cycle 1 Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 7
ng*h/mL | 2795.782 (35.7) | 3393.296 (30.4)

6. Primary Outcome: Summary of Nilotinib Steady-state PK Parameters: AUCss
Description: The steady-state PK profiles of nilotinib in pediatric patients were estimated using trough sampling following multiple 230 mg/m2 bid doses
Time Frame: Cycle 1 Day 8 - Cycle 1 Day 28
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 7
ng*h/mL | 15129.182 (38.0) | 14383.076 (33.6)

7. Primary Outcome: Summary of Nilotinib Steady-state PK Parameters: CLF (Body Surface Area (BSA) Adjusted)
Description: as for outcome 6
Time Frame: Cycle 1 Day 8 - Cycle 1 day 28
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/m^2)
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 7
L/h/m^2) | 15.356 (38.7) | 15.922 (37.0)

8. Primary Outcome: Summary of Nilotinib Steady-state PK Parameters: Cmin
Description: The full PK profiles of nilotinib in pediatric patients were assessed using serial sampling following a single 230 mg/m2 dose.
Time Frame: Cycle 1 Day 8 - Cycle 1 Day 28
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 7
ng/mL | 804.791 (33.7) | 1072.850 (20.5)

9. Secondary Outcome: Number of Ph+ CML Participants With Cytogenic Response
Description: Cytogenetic response was initially assessed as the percentage of Ph+ metaphases in the bone marrow (BM) and performed within 21 days prior to study entry. A major cytogenetic response (0% to 35% Ph+ metaphases test positive for the Philadelphia chromosome) combines both complete cytogenetic (CCyR) and partial cytogenetic response (PCyR). CCyR implies 0% Ph+ metaphases in the BM, PCyR is > 0% to 35%, minor cytogenetic response (mCyR) is > 35% to 65%, minimal response is > 65% to 95% and no response is > 95% Ph+ metaphases in the BM.
Time Frame: minimum of 12 cycles (28 days per cycle)
Population: FAS consist of all patients (pts) who passed screening & are enrolled into study. Patients may or may not have taken study drug. One (1) Ph+ CML patient in Group 2 was Ph+ at baseline & discontinued study prior to subsequent cytogenetic assessment. This pt doesn't appear in any cytogenic response category.
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 6
Participants
  Complete cytogenic response (CCyR) | 2 | 2
  Partial cytogenic response (PCyR) | 0 | 1
  Minor cytogenic response (mCyR) | 0 | 1
  Minimal | 0 | 0
  None | 0 | 0
  Absence of Ph+ at baseline | 3 | 1

10. Secondary Outcome: Number of Ph+ CML Participants With Major Molecular Response (MMR)
Description: The bcr-abl gene fusion encodes for a BCR-ABL fusion protein. Depending on the precise location of the fusion, the molecular weight of this protein can range from 185 to 210 kDa. Consequently BCR-ABL is referred to as p185 or p210 transcript. For the patients expressing the major BCR-ABL transcript p210, molecular response was defined and reported as the percent ratio of BCR-ABL transcripts/control gene transcripts converted to a reference standard according to the International Scale (IS). A major molecular response (MMR) is defined as a BCR-ABL/control gene ratio ≤ 0.1% (equal to a 3 log reduction in BCR-ABL transcripts) on the IS. In this study, the control gene was abl.
Time Frame: minimum of 12 cycles (28 days per cycle)
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 6
Participants
  Yes | 1 | 2
  No | 4 | 4

11. Secondary Outcome: Efficacy Endpoints for Ph+ ALL Patients
Description: Best Response in Ph+ ALL patients was defined as either Complete Remission (CR) with platelet recovery, Complete Remission (CR) with incomplete platelet recovery, Partial Remission (PR) or Stable disease. Stable disease was defined is defined as failure to qualify for either CR, PR, or progressive disease.
Time Frame: minimum of 12 cycles (28 days per cycle)
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 3 | 1
Participants
  Complete Remission with platelet recovery | 2 | 1
  Complete Remission w/incomplete platelet recovery | 0 | 0
  Partial remission | 0 | 0
  Stable disease | 1 | 0
  Progressive disease | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 2/8 | 3/7
Other Adverse Events (participants affected / at risk) | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=8) | Group 2 (N=7)
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Appendix disorder (Gastrointestinal disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=8) | Group 2 (N=7)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 3
Odynophagia (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 0 | 1
Catheter site pain (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Xerosis (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2
Bronchitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 2
Fungal skin infection (Infections and infestations) | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0
Lip infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 3 | 1
Skin infection (Infections and infestations) | 0 | 2
Tinea pedis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Bilirubin conjugated increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 3
Blood bilirubin unconjugated increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2
Blood phosphorus decreased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 0 | 2
Blood uric acid increased (Investigations) | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Headache (Nervous system disorders) | 4 | 2
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.